CLINICAL TRIAL: NCT06375499
Title: Comparison of the Performance and Safety of T2769 Versus Hylo-Forte® in the Treatment of Moderate to Severe Dry Eye Syndrome.
Brief Title: Performance and Safety of T2769 Versus Hylo-Forte® in the Treatment of Moderate to Severe Dry Eye Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2769-004
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Results first posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2769 (Experimental): Hyaluronic acid, Trehalose, Naaga
  Route of administration: topical, ocular use
  Interventions: Device: T2769
- Hylo-Forte® (Active Comparator): Hyaluronic acid
  Route of administration: topical, ocular use
  Interventions: Device: Hylo-Forte®

INTERVENTIONS:
Device: T2769 — Daily dose regimen: 1 drop in each eye, from 3 to 6 times daily.
  Arms: T2769
Device: Hylo-Forte® — Daily dose regimen: 1 drop in each eye, from 3 to 6 times daily.
  Arms: Hylo-Forte®

SUMMARY:
The objective is to demonstrate the non-inferiority of T2769 compared to Hylo-Forte® in terms of the change from baseline (D1) in total ocular surface staining score assessed on Oxford 0-15 scale, in the study eye at the D36 visit.

The investigation is defined as a post-market stage. The clinical investigation design is confirmatory.

ELIGIBILITY:
Main Inclusion Criteria (At Screening visit):

* Informed consent signed and dated (obtained prior to initiating any procedures).
* Patient aged ≥18 years old.
* Persistence of dry eye syndrome, despite artificial tears use in the previous month prior to the screening visit

Main Exclusion Criteria (At both Screening and Randomisation visits):

* Far Best-Corrected Visual Acuity (BCVA) ≥+0.7 LogMar (e.g., ≤0.2 in decimal value or ≤20/100 Snellen equivalent or ≤50 letters Early Treatment Diabetic Retinopathy Study (ETDRS)).
* Patient with previous or current ophthalmic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Czechia (2):
  - OFTEX, s.r.o., Prague
  - Axon Clinical, s.r.o., Prague
- Hungary (2):
  - Ganglion Medical Center, Pécs, Baranya
  - Ermellek Egeszsegcentrum, Létavértes, Hb

RESULTS

PARTICIPANT FLOW:
Groups:
- T2769: T2769 (Thealoz® Total) T2769 is a sterile, phosphate-free and pH neutral solution. It contains Trehalose, Sodium Hyaluronate (SH) and Naaga.
- Hylo-Forte: HYLO-FORTE® is a sterile, phosphate and preservative-free solution for ocular use containing sodium hyaluronate, citric acid anhydrous, sodium citrate and sorbitol.
Period: Overall Study
Arm/Group | T2769 | Hylo-Forte
Started | 36 | 38
Completed | 35 | 38
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- T2769: Test device: T2769 (Thealoz® Total) T2769 is a sterile, phosphate-free and pH neutral solution. It contains Trehalose, Sodium Hyaluronate (SH) and Naaga.
- Total: Total of all reporting groups
Arm/Group | T2769 | Hylo-Forte | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.42) | 47.5 (14.44) | 50.6 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 30 | 35 | 65
  Czechia | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate the Non-inferiority of T2769 Compared to Hylo-Forte® in Terms of Total Ocular Surface Staining (Oxford Score).
Description: The primary endpoint is the change from baseline (Day 1) in total ocular surface staining grade according to Oxford Scale 0-15 grading scheme at D36 in the study eye. Minimum value is 0 (better case) and maximum value is 15 (worse case)
Time Frame: Oxford 0-15 grading scheme: is assessed at Day 1, Day 15 and Day 36
Population: Day 1-Baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- T2769: Test device: T2769 (Thealoz® Total)
- Hylo-Forte: Comparator: HYLO-FORTE®
Arm/Group | T2769 | Hylo-Forte
Number analyzed (Participants) | 35 | 38
score on a scale | -1.3 [-2.0 to -0.5] | -1.2 [-1.9 to -0.5]

ADVERSE EVENTS:
Time Frame: 7 weeks from D-10 to D36 (+3 days)
Description: AE: Any untoward medical occurrence, unintended disease or injury or untoward clinical signs in subjects, users or other persons whether or not related to IMD.
  This includes events related to IMD or comparator, events related to the procedures involved, For users or other persons, this definition is restricted to events related to use of the IMD or comparator.
  Adverse event is an incident. REPORTING: Any incident must report to Sponsor within 24 hours of awareness using incident form.
Arm/Group | T2769 | Hylo-Forte
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT06375499/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT06375499/SAP_001.pdf